CLINICAL TRIAL: NCT01867567
Title: Early Bandage Removal Post-Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Principal Investigator, David Peleg, Staff Physician, Ziv Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CSBandage
Record Dates: First submitted 2013-05-26; First posted 2013-06-04 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Wound Disruption; Wound Infection
Keywords: cesarean; bandage removal; infection; disruption; satisfaction; patient satisfaction
MeSH Terms: conditions — Wound Infection; Infections; Personal Satisfaction; Patient Satisfaction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 6 Hours (Experimental): Removal of bandage after 6 hours
  Interventions: Procedure: abdominal bandage
- 24 hours (Active Comparator): removal of bandage after 24 hours
  Interventions: Procedure: abdominal bandage

INTERVENTIONS:
Procedure: abdominal bandage

SUMMARY:
Women undergoing their first second or third cesarean section will be randomized into two groups. One group will have the abdominal bandage removed at 6 hours post-surgery and the other group will have the bandage removed at 24 hours. Staple removal will be at 5 - 7 days for both groups. The incision will be inspected at the time of staple removal. The 2 groups will be compared for incision disruption and infection. Also, the women will be asked about their satisfaction for time of bandage removal.

ELIGIBILITY:
Inclusion Criteria:

* age of 18 to 44
* elective cesarean section, primary or repeat
* low risk pregnancy

Exclusion Criteria:

* under the age of 18 and above the age of 44
* diabetes, preeclampsia or other pregnancy complications
* unable or unwilling to give informed consent
* chorioamnionitis
* BMI over 35
* more than 3 cesareans

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 320 (Actual)
Dates: Start 2013-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Wound Disruption | 5 - 7 days

SECONDARY OUTCOMES:
Wound Infection | 5 - 7 days
Patient satisfaction | 5 - 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- Ziv Medical center, Safed, Israel